CLINICAL TRIAL: NCT03417752
Title: Unlocking the Potential of VA Means Safety Programs: An Examination of the Use of Public Messaging for the Promotion of Firearm Safety to Veterans
Brief Title: The Use of Public Messaging for the Promotion of Firearm Safety to Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Karras, Health Science Specialist, Canandaigua VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 910434
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure to firearm safety Public Service Announcement (PSA) (Experimental): Exposure to the firearm safety PSA (approx. 2.5 minutes long) once per week for 3 weeks.
  Interventions: Other: Exposure to firearm safety PSA
- Exposure to a mix of PSAs (Experimental): Exposure to a general health promotion video (approx. 2 minutes long) 1 week post-randomization followed by exposure to firearm safety PSA at 2- and 3-weeks post-randomization.
  Interventions: Other: Exposure to firearm safety PSA; Other: Exposure to health promotion PSA
- Active control (Active Comparator): Exposure to the general health promotion video once per week for 3 weeks.
  Interventions: Other: Exposure to health promotion PSA

INTERVENTIONS:
Other: Exposure to firearm safety PSA — Exposed to firearm safety PSA
  Arms: Exposure to a mix of PSAs; Exposure to firearm safety Public Service Announcement (PSA)
Other: Exposure to health promotion PSA — Exposed to general health promotion PSA
  Arms: Active control; Exposure to a mix of PSAs

SUMMARY:
This pilot study seeks to determine if exposure to the firearm safety public service announcement (PSA) developed by the U.S. Department of Veterans Affairs (VA) is associated with changes in related beliefs and safe storage practices. Participants are randomly assigned to message exposure or control conditions. Data from this project will inform injury prevention outreach efforts targeted towards Veteran populations.

ELIGIBILITY:
Inclusion Criteria:

* Veterans of all gender/sex, race/ethnicities
* Living in United States
* Fluent in English language
* Capable of understanding the goals of the study
* Possess computer/internet access

Exclusion Criteria:

* Not a U.S. Veteran living in the United States
* Determined to be cognitively impaired
* Currently institutionalized (e.g., hospitalized; incarcerated, etc.)
* Do not possess computer/internet access

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Karras, PhD, Principal Investigator — VA Center of Excellence for Suicide Prevention

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exposure to Firearm Safety PSA: Exposure to the firearm safety PSA (approx. 2.5 minutes long) once per week for 3 weeks.
  Exposure to firearm safety PSA: Exposed to firearm safety PSA
Period: Overall Study
Arm/Group | Exposure to Firearm Safety PSA | Exposure to a Mix of PSAs | Active Control
Started | 149 | 175 | 150
Completed | 115 | 133 | 110
Not Completed | 34 | 42 | 40

BASELINE CHARACTERISTICS:
Population: analysis restricted to participants with baseline and exit responses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposure to Firearm Safety Public Service Announcement (PSA) | Exposure to a Mix of PSAs | Active Control | Total
Number analyzed (Participants) | 115 | 133 | 110 | 358
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-59 yrs old | 50 | 58 | 48 | 156
  Age: 60-69 yrs old | 29 | 33 | 28 | 90
  Age: 70+ years old | 36 | 42 | 34 | 112
Sex/Gender, Customized [Count of Participants; unit: Participants]
  male | 104 | 120 | 99 | 323
  female | 11 | 13 | 11 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race: white | 97 | 113 | 92 | 302
  race: Non-white | 18 | 20 | 18 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported Injury Prevention Belief
Description: Number of participants with self-reported response to belief that "safe storage of household firearms is effective for reducing injury or death."
Time Frame: baseline
Population: Analyses were restricted to participants that completed both baseline and exit surveys. Descriptive statistics were tabulated by frequencies and weighted percentages or mean and standard deviation, as appropriate.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure to Firearm Safety PSA | Exposure to a Mix of PSAs | Active Control
Number analyzed (Participants) | 115 | 133 | 110
Participants
  Agree | 66 | 73 | 57
  Disagree | 49 | 60 | 53

2. Primary Outcome: Number of Participants With Self-reported Injury Prevention Belief
Description: as for outcome 1
Time Frame: 3 weeks post-baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure to Firearm Safety PSA | Exposure to a Mix of PSAs | Active Control
Number analyzed (Participants) | 115 | 133 | 110
Participants
  Agree | 71 | 79 | 64
  Disagree | 44 | 54 | 46

3. Secondary Outcome: Number of Participants Who Self-reported Firearm Storage Behavior at Baseline
Description: Number of participants at baseline with self-reported safe household firearm storage (restricted to participants with self-reported firearm access)
Time Frame: baseline
Population: Analyses were restricted to participants that reported firearm access. Descriptive statistics were tabulated by frequencies and weighted percentages or mean and standard deviation, as appropriate.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure to Firearm Safety PSA | Exposure to a Mix of PSAs | Active Control
Number analyzed (Participants) | 64 | 71 | 60
Participants
  Safe storage (yes) | 8 | 23 | 24
  safe storage (no) | 56 | 48 | 36

4. Secondary Outcome: Number of Participants Who Self-reported Firearm Storage Behavior at Exit
Description: Number of participants at exit with self-reported safe household firearm storage (restricted to participants with self-reported firearm access)
Time Frame: 3 weeks post-baseline
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Exposure to Firearm Safety PSA | Exposure to a Mix of PSAs | Active Control
Number analyzed (Participants) | 64 | 71 | 60
Participants
  safely stored (yes) | 7 | 25 | 23
  safely stored (no) | 57 | 46 | 37

ADVERSE EVENTS:
Time Frame: over 1 calendar year
Description: Adverse and serious adverse events were defined using standard definitions.
Arm/Group | Exposure to Firearm Safety PSA | Exposure to a Mix of PSAs | Active Control
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/133 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/133 | 0/110
Other Adverse Events (participants affected / at risk) | 0/115 | 0/133 | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03417752/Prot_SAP_000.pdf